CLINICAL TRIAL: NCT04354415
Title: Comparing Open Carpal Tunnel or Trigger Finger Release Procedures Performed Under Local Anesthesia With or Without the Use of a Tourniquet: A Randomized Controlled Trial
Brief Title: Tourniquet vs. No Tourniquet for Carpal Tunnel and Trigger Finger Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Eli Saleh, Plastic Surgery Resident, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-CEMTL(6518)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Carpal Tunnel Syndrome; Trigger Finger
Keywords: Tourniquet; WALANT; Patient-Centered
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: This was a randomized controlled trial comparing patients undergoing open carpal tunnel or trigger finger release with or without the use of a tourniquet. This was an equivalence trial in terms of operative time, bleeding scores and peri-operative complication rates. In addition, peri-operative subjective patient experience was investigated for both techniques. This was measured based on a numerical rating scale (NRS) for pain, anxiety and overall satisfaction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet Group (Active Comparator): Tourniquet application during procedures
  Interventions: Procedure: Carpal tunnel or trigger finger release
- Non-Tourniquet group (Experimental): No application of tourniquet for procedures
  Interventions: Procedure: Carpal tunnel or trigger finger release

INTERVENTIONS:
Procedure: Carpal tunnel or trigger finger release — Carpal tunnel or trigger finger release with and without the use of tourniquet

SUMMARY:
Background: Trigger finger and carpal tunnel syndrome are two of the most common conditions treated by the hand surgeon. During these procedures, a tourniquet is often used to minimize bleeding and improve visualization of the operative field. However, it may be associated with pain and discomfort. To date, there are few prospective studies investigating the safety and outcomes of tourniquet-free minor hand procedures.

Methods: This is a randomized controlled trial comparing patients undergoing open carpal tunnel or trigger finger release with or without the use of a tourniquet. This is an equivalence trial in terms of operative time, bleeding scores and peri-operative complication rates. In addition, peri-operative subjective patient experience will be investigated for both techniques. This will be measured based on a numerical rating scale (NRS) for pain, anxiety and overall satisfaction. The primary goal of this study is to to determine the efficacy and patient preference of the the differing techniques.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing patients undergoing open carpal tunnel or trigger finger release with or without the use of a tourniquet. This will be a parallel study by design where the allocation ratio between the two groups will be set to be 1:1.

Patients are to be recruited on the day of the procedure. Upon arrival, they will be presented with the research project and given the information pamphlet and consent forms. Sufficient time to read these documents will be allocated.

For the purpose of this RCT, the same volume and concentration of the solution will be injected in the surgical site prior to entering the operating room, thereby allowing epinephrine to full take effect. The solution used by the hand surgeons will include 8 cc of 2% xylocaine with epinephrine mixed with 3 cc of 0.5% Marcaine with epinephrine. Eight millilitres will be used for the CT releases and 4 millilitres for the TF releases. Once in the room, the patient's arm will be disinfected and draped in a similar fashion, and surgery will proceed without inflation of the tourniquet. A system will be implemented so that before patient A's surgery begins, patient B will be injected in a separate room. By the time patient B's surgery begins, a minimum of 30 minutes will have elapsed since his injection. Other than the differences in tourniquet use, all other procedure-specific elements will be identical, namely the size and location of the incision, the surgical technique, skin closure, type of dressing, rehabilitation and post-operative follow-up.

The primary outcome of interest is peri-operative patient experience. The aim is to demonstrate the superiority of the no tourniquet technique with respect to the patients' subjective experience peri-operatively. This will be measured based on a numerical rating scale (NRS) for pain, anxiety and overall satisfaction. As secondary outcomes, operative time, bleeding control and short-term complication rates will be looked at and compared between the two groups.

To achieve statistical significance, at least 31 patients will be needed in each group to show a minimal decrease of 33% on the NRS scales evaluation of the postoperative pain and overall experience with an α error of 0,05 and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have been over the age of 18 at the time of surgery
2. must have had either an electromyographically confirmed CTS and/or a clinically significant triggering or locking digit.
3. Patients must have been able to understand and complete the pre-and post-operative questionnaires which were administered in either English or French.

Exclusion Criteria:

1. contra-indications for subcutaneous epinephrine use
2. history of digital gangrene
3. buerger's disease
4. previous replantation
5. Raynaud
6. Sclerodactyly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Peri-operative patient experience | In the immediate post-operative period
  Based on Numerical rating scale (NRS) from 1 to 10. 1 being no pain at all, 10 being unbearable pain throughout procedure and post-operatively

SECONDARY OUTCOMES:
Operative time | Assessed in the immediate post-operative period
  time from beginning to end of surgery
Bleeding levels | Assessed peri-operatively and noted in the immediate post-operative period
  3-point ordinal scale:
  1. No bleeding
  2. minor bleeding controlled with dabbing
  3. bleeding requiring use of electrocautery
Peri-operative complication | In the immediate post-operative period
  Peri-operative complications including nerve or tendon damage
Post-operative complications | 1 week
  Hematoma, infection and wound dehiscence/breakdown

CONTACTS AND LOCATIONS:
Overall Officials: Dominique M Tremblay, MD, Principal Investigator — Université de Montréal (Hospital Maisonneuve-Rosemont)
Locations (1):
- Hospital Maisonneuve Rosemont, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No